CLINICAL TRIAL: NCT00848926
Title: A Pivotal Study of SGN-35 in Treatment of Patients With Relapsed or Refractory Hodgkin Lymphoma (HL)
Brief Title: A Pivotal Open-Label Trial of Brentuximab Vedotin for Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG035-0003; 2008-006034-10 (EudraCT Number)
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2015-06

CONDITIONS: Disease, Hodgkin
Keywords: Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Disease, Hodgkin; Hematologic Diseases; Lymphoma; monomethylauristatin E; Drug Therapy; Immunotherapy
MeSH Terms: conditions — Hodgkin Disease; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brentuximab vedotin (Experimental)
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg every 3 weeks by intravenous infusion
  Other Names: SGN-35; ADCETRIS

SUMMARY:
This is a single-arm, open-label, multicenter, pivotal clinical trial to evaluate the efficacy and safety of brentuximab vedotin (SGN-35) as a single agent in patients with relapsed or refractory Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory Hodgkin lymphoma who have previously received autologous stem cell transplant.
* Histologically confirmed CD30-positive disease; tissue from the most recent post diagnostic biopsy of relapsed/refractory disease must be available for confirmation of CD30 expression via slides or tumor block.
* Fluorodeoxyglucose-avid disease by positron emission tomography and measurable disease of at least 1.5 cm as documented by spiral computed tomography.
* At US sites patients greater than or equal to 12 years of age may be enrolled. At non-US sites patients must be greater than or equal to 18 years of age.

Exclusion Criteria:

* Previous treatment with brentuximab vedotin.
* Previously received an allogeneic transplant.
* Congestive heart failure, Class III or IV, by the New York Heart Association criteria.
* History of another primary malignancy that has not been in remission for at least 3 years.
* Known cerebral/meningeal disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Fong, MD, PhD, Study Director — Seagen Inc.
Locations (27):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of California at Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Loyola University Medical Center Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Baylor Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- Belgium (2):
  - UZ Gasthuisberg, Leuven
  - Cliniques Universitaires UCL de Mont-Goddine, Yvoir
- Canada (2):
  - B.C Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
- France (3):
  - Institut Paoli Calmettes, Marseille
  - Hospital Saint Louis, Paris
  - Centre Henri Becquerel, Rouen
- Instituto di Ematologia ed Oncologia Medica, Bologna, Italy

REFERENCES:
- [Result] Younes A, Gopal AK, Smith SE, Ansell SM, Rosenblatt JD, Savage KJ, Ramchandren R, Bartlett NL, Cheson BD, de Vos S, Forero-Torres A, Moskowitz CH, Connors JM, Engert A, Larsen EK, Kennedy DA, Sievers EL, Chen R. Results of a pivotal phase II study of brentuximab vedotin for patients with relapsed or refractory Hodgkin's lymphoma. J Clin Oncol. 2012 Jun 20;30(18):2183-9. doi: 10.1200/JCO.2011.38.0410. Epub 2012 Mar 26. PMID 22454421
- [Derived] Chen R, Gopal AK, Smith SE, Ansell SM, Rosenblatt JD, Savage KJ, Connors JM, Engert A, Larsen EK, Huebner D, Fong A, Younes A. Five-year survival and durability results of brentuximab vedotin in patients with relapsed or refractory Hodgkin lymphoma. Blood. 2016 Sep 22;128(12):1562-6. doi: 10.1182/blood-2016-02-699850. Epub 2016 Jul 18. PMID 27432875
- [Derived] Gopal AK, Chen R, Smith SE, Ansell SM, Rosenblatt JD, Savage KJ, Connors JM, Engert A, Larsen EK, Chi X, Sievers EL, Younes A. Durable remissions in a pivotal phase 2 study of brentuximab vedotin in relapsed or refractory Hodgkin lymphoma. Blood. 2015 Feb 19;125(8):1236-43. doi: 10.1182/blood-2014-08-595801. Epub 2014 Dec 22. PMID 25533035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: Feb 2009 - Aug 2009
Groups:
- Brentuximab Vedotin: Brentuximab vedotin 1.8 mg/kg every 3 weeks by intravenous (IV) infusion
Period: Treatment Period
Arm/Group | Brentuximab Vedotin
Started | 102
Completed | 18 (Number who completed 16 cycles of treatment)
Not Completed | 84
Not completed — Progressive disease | 45
Not completed — Adverse Event | 20
Not completed — Physician Decision | 12
Not completed — Withdrawal by Subject | 7
Period: Follow-up Period
Arm/Group | Brentuximab Vedotin
Started | 102 (All participants were to be followed after treatment)
Completed | 90 (Completed survival follow-up due to death [57] or study termination by sponsor [33])
Not Completed | 12
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- Brentuximab Vedotin: Brentuximab vedotin 1.8 mg/kg every 3 weeks by IV infusion
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
Age, Customized [Median (Full Range); unit: years] | 31.0 [15 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 89
  More than one race | 0
  Unknown or Not Reported | 1
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — 0 = Normal activity
  1. = Symptoms but ambulatory
  2. = In bed <50% of the time
  3. = In bed >50% of the time
  4. = 100% bedridden
  5. = Dead
  participants
    0 | 42
    1 | 60
    2-5 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate by Independent Review Group
Description: Percentage of participants who achieved a best response of complete remission (CR, disappearance of all evidence of disease) or partial remission (PR, regression of greater than or equal to 50% of measurable disease and no new sites) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: up to 12 months
Population: Intention to treat
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
percent of participants | 75 [64.9 to 82.6]

2. Secondary Outcome: Complete Remission Rate by Independent Review Group
Description: Percentage of participants who achieved a best response of CR (disappearance of all evidence of disease) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: up to 12 months
Population: Intention to treat
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
percent of participants | 33 [24.3 to 43.4]

3. Secondary Outcome: Duration of Objective Response by Kaplan-Meier Analysis
Description: Duration of objective response (CR + PR) by independent review group, defined as time of initial response until disease progression or death.
Time Frame: up to approximately 4 years
Population: Participants with objective response among the intention to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 76
months | 6.7 [3.6 to 14.8]

4. Secondary Outcome: Duration of Objective Response in Participants With Complete Remission by Kaplan-Meier Analysis
Description: Duration of response from start of first objective tumor response (CR or PR) by independent review group to disease progression or death due to any cause in participants with CR.
Time Frame: up to approximately 4 years
Population: Participants with complete remission among the intention to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 34
months | 27.9 [10.8 to NA] — Insufficient number of events to estimate upper bound

5. Secondary Outcome: Progression-free Survival by Kaplan-Meier Analysis
Description: Time from start of study treatment to disease progression per independent review group or death due to any cause.
Time Frame: up to approximately 4 years
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
months | 5.6 [5.0 to 9.0]

6. Secondary Outcome: Overall Survival
Description: Time from start of study treatment to date of death due to any cause.
Time Frame: up to approximately 6 years
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
months | 40.5 [28.7 to 61.9]

7. Secondary Outcome: Adverse Events by Severity, Seriousness, and Relationship to Treatment
Description: Counts of participants who had adverse events or treatment-emergent adverse events (TEAE, defined as newly occurring or worsening after first dose). Serious adverse events are reported from the time of informed consent. National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 3.0) were used to assess severity (1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death). Relatedness to study drug was assessed by the investigator (Yes/No). Participants with multiple occurrences of an adverse event within a category are counted once within the category.
Time Frame: up to 12 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
participants
  Any TEAE | 100
  TEAE related to study drug | 94
  TEAE with severity grade >/=3 | 56
  Serious adverse event | 25
  Serious adverse event related to study drug | 14
  Discontinued treatment due to adverse event | 20

8. Secondary Outcome: Hematology Laboratory Abnormalities >/= Grade 3
Description: Counts of study participants with post-baseline hematology laboratory abnormalities of Grade 3 or greater per NCI CTCAE version 3.0. Participants with multiple occurrences of a laboratory abnormality within a category are counted once in that category.
Time Frame: up to 12 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
participants
  Any >/= Grade 3 hematology laboratory abnormality | 35
  Hemoglobin (low) | 7
  Leukocytes (low) | 6
  Lymphocytes (low) | 20
  Neutrophils (low) | 12
  Platelets (low) | 7

9. Secondary Outcome: Chemistry Laboratory Abnormalities >/= Grade 3
Description: Counts of study participants with post-baseline chemistry laboratory abnormalities of Grade 3 or greater per NCI CTCAE version 3.0. Participants with multiple occurrences of a laboratory abnormality within a category are counted once in that category.
Time Frame: up to 12 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
participants
  Any >/= Grade 3 chemistry laboratory abnormality | 14
  Alanine aminotransferase (high) | 1
  Albumin (low) | 1
  Calcium (low) | 1
  Glucose (high) | 7
  Potassium (low) | 2
  Sodium (high) | 1
  Urate (high) | 1

10. Secondary Outcome: Area Under the Curve
Description: Area under the serum concentration-time curve from time 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All participants who received treatment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day * microgram/mL
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
day * microgram/mL | 88 (46)

11. Other Pre Specified Outcome: B Symptom Resolution
Description: Percentage of participants with lymphoma-related symptoms (B symptoms: fever, night sweats, or weight loss >10%) at baseline who achieved resolution of all B symptoms at any time during the treatment period.
Time Frame: up to 12 months
Population: Participants with B symptoms at baseline
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 35
percent of participants | 77 [59.9 to 89.6]

12. Secondary Outcome: Maximum Serum Concentration
Description: Maximum serum concentration from 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All participants who received treatment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
microgram/mL | 35 (17)

13. Secondary Outcome: Time of Maximum Serum Concentration
Description: Time of maximum serum concentration from 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All participants who received treatment
Measure: Median (Full Range); unit: days
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 102
days | 0.02 [0.02 to 0.02]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events through 30 days after last dose (up to 12 months)
Arm/Group | Brentuximab Vedotin
Serious Adverse Events (participants affected / at risk) | 25/102
Other Adverse Events (participants affected / at risk) | 97/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=102)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Demyelinating polyneuropathy (Nervous system disorders) | 2
Diabetic coma (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=102)
Anaemia (Blood and lymphatic system disorders) | 9
Lymphadenopathy (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 37
Nausea (Gastrointestinal disorders) | 43
Vomiting (Gastrointestinal disorders) | 22
Chills (General disorders) | 13
Fatigue (General disorders) | 47
Pain (General disorders) | 7
Pyrexia (General disorders) | 30
Bronchitis (Infections and infestations) | 8
Herpes zoster (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 38
Urinary tract infection (Infections and infestations) | 6
Weight decrease (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 19
Peripheral motor neuropathy (Nervous system disorders) | 11
Peripheral sensory neuropathy (Nervous system disorders) | 48
Anxiety (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less